CLINICAL TRIAL: NCT05490615
Title: Virtual Mindfulness for Autistic Adults: A Randomized Controlled Trial
Brief Title: The Virtual Mindfulness Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Yona Lunsky, Professor, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Record Dates: First submitted 2022-08-04; First posted 2022-08-05 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Autism
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness Intervention (Group-A) (Experimental): Total length of study for participants in Group-A:15 Week
  Six weekly sessions (each 60 minutes in length) of group based virtual mindfulness instruction, co-led by a mindfulness teacher and two autistic adults, following a workbook designed for autistic adults. In between sessions, participants are encouraged to complete homework and keep a record of when they practice formal and informal mindfulness practices. In addition, participants are provided with a link to autism informed mental health resources (https://www.yorku.ca/health/lab/ddmh/am-help/)
  Interventions: Behavioral: Virtual Mindfulness
- Waitlist Control (Group-B) (No Intervention): Total length of study for participants in Group-B: 30 Week
  A waitlist control group is an ethical alternative to no-treatment control groups when studying psychological and behavioral interventions. This group will have access to intervention at the end of the study as well. All waitlist participants are provided with a link to autism informed mental health resources (https://www.yorku.ca/health/lab/ddmh/am-help/)

INTERVENTIONS:
Behavioral: Virtual Mindfulness — Investigators have previously developed and tested a virtual mindfulness program. Six 1-hour weekly group sessions will be led on WebEx. Focus will be on skill building through the teaching of formal and informal mindfulness practices. The intervention, based on the MBSR curriculum, has been modified to make it more accessible for autistic adults. The curriculum developed for this program was designed with autistic advisors guiding the team on the length of meditations, the language used when giving instructions, and the range of techniques that would be most helpful for autistic adults. Each activity is presented as optional, recognizing that some people may find certain silent sensory experiences too distressing. Autistic advisors will participate in sessions as co-facilitators and multiple communication options will be available to group participants (text and audio, camera on or off).
  Arms: Mindfulness Intervention (Group-A)

SUMMARY:
The purpose of this study is to test the effectiveness of a virtual group mindfulness intervention for autistic adults on their mental health and well-being, compared to a group who has not received the virtual group intervention. Specifically, the investigators will compare change across multiple indicators of mental health and well-being for participants, post-intervention, and at 15 weeks follow-up, to participants in a waitlist control group who have not yet received the intervention.

DETAILED DESCRIPTION:
It is well recognized that autistic individuals experience high rates of mental health issues, but that needed mental health services are often inaccessible. There is some evidence to suggest that mindfulness-based therapies may help to reduce some of these challenges for autistic adults. While in person interventions may be helpful, there are also benefits to participating in virtually based interventions, particularly during the pandemic. Virtual groups have the added benefit of not requiring travel for people who have difficulties with travel because of anxiety or financial constraints. For some autistic individuals, virtual engagement can be preferred over in person interactions because of the flexibility that virtual interactions allow (camera on or off, communicating with text or speaking, being able to attend from home in a familiar and comfortable space).

In a prior CAMH led study, the investigators demonstrated that autism-informed adaptations to a standard mindfulness-based virtually delivered group intervention led to self-reported improvements in mindfulness, self-compassion, and distress, with changes maintained at three months follow-up. This prior study lacked a control group, however so it is not known whether the positive impacts reported were specific to the mindfulness-based intervention itself or to other factors. Building on this previous work, there is a need to study whether improvements are also evident when compared to individuals who do not take part in the intervention.

The purpose of this study is to test the effectiveness of a virtual group mindfulness intervention for autistic adults on their mental health and well-being, compared to a group who has not received the virtual group intervention. Specifically, the investigators will compare change across multiple indicators of mental health and well-being for participants, post-intervention, and at 15 weeks follow-up, to participants in a waitlist control group who have not yet received the intervention.

Study Design: Randomized controlled trial with waitlist control.

Hypotheses We expect that participants in the mindfulness-based intervention group will report improvements in self-reported distress (primary outcome), mindfulness, self-compassion, and sense of autistic belonging (secondary outcomes), relative to the waitlist control group, which will be maintained at 15 weeks follow-up.

Survey Evaluation: All participants will provide pre, post and follow-up survey data related to either a 6-week virtual mindfulness course or waitlist. Participants will fill out survey measures evaluating the impact of either the intervention or waitlist on distress levels, self-compassion, mindfulness, and connections from baseline (Time 1) to week 7 (Time 2) and week 15 (Time 3). In addition, the waitlist control group (Group B) will be offered virtual mindfulness intervention from week 16 to week 21 and will be asked to complete 2 additional set of questionnaires at week 22 and at week 30, thus providing data pre and post with follow-up related to the mindfulness intervention.

Study Setting: This study will be delivered virtually but will be offered through CAMH, Toronto.

Target Population We aim to recruit in total 80 autistic adults from across Canada.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years and older;
* Autistic
* Proficient in English;
* Able to independently complete survey questionnaires;
* Able to independently participate in an online based group;
* Access to internet and computer/tablet

Exclusion Criteria:

* Presence of intellectual disability;
* Unable to comprehend English or speak or write in English;
* No access to internet and computer/tablet.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2022-11-17 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
Psychological distress: measured using the Depression and Anxiety Stress Scale (DASS-21) | Baseline or enrolment (Group-A and Group B)
  To assess psychological distress, including a 7-item depression subscale, a 7 -item anxiety subscale, and a 7-item stress subscale, each on a 4-point Likert scale, with higher scores indicating higher levels of distress. Total scores for each subscale range from 0 to 42 (summed numbers in each subscale multiplied by 2).
Psychological distress: measured using the Depression and Anxiety Stress Scale (DASS-21) | 7 Weeks (Group-A and Group B)
  To assess psychological distress, including a 7-item depression subscale, a 7 -item anxiety subscale, and a 7-item stress subscale, each on a 4-point Likert scale, with higher scores indicating higher levels of distress. Total scores for each subscale range from 0 to 42 (summed numbers in each subscale multiplied by 2).
Psychological distress: measured using the Depression and Anxiety Stress Scale (DASS-21) | 15 Weeks (Group-A and Group B)
  To assess psychological distress, including a 7-item depression subscale, a 7 -item anxiety subscale, and a 7-item stress subscale, each on a 4-point Likert scale, with higher scores indicating higher levels of distress. Total scores for each subscale range from 0 to 42 (summed numbers in each subscale multiplied by 2).
Psychological distress: measured using the Depression and Anxiety Stress Scale (DASS-21) | 22 Weeks (Group-B)
  To assess psychological distress, including a 7-item depression subscale, a 7 -item anxiety subscale, and a 7-item stress subscale, each on a 4-point Likert scale, with higher scores indicating higher levels of distress. Total scores for each subscale range from 0 to 42 (summed numbers in each subscale multiplied by 2).
Psychological distress: measured using the Depression and Anxiety Stress Scale (DASS-21) | 30 Weeks (Group-B)
  To assess psychological distress, including a 7-item depression subscale, a 7 -item anxiety subscale, and a 7-item stress subscale, each on a 4-point Likert scale, with higher scores indicating higher levels of distress. Total scores for each subscale range from 0 to 42 (summed numbers in each suscale multiplied by 2).

SECONDARY OUTCOMES:
Autistic Participant Self Compassion - measured using Self Compassion Scale-Short Form (SCS-SF) | Baseline/enrolment (Group-A and Group B)
  12-item measure that assesses the ability to demonstrate care and kindness toward oneself, and acceptance of one's own imperfections. Self-compassion is often a focus of mindfulness-based interventions because of the interrelatedness with state mindfulness. Responses will be given using a 5-point Likert scale that ranged from 1 ("Almost never") to 5 ("Almost always"), yielding a total score between 12 and 60, with higher scores indicating greater self-compassion.
Autistic Participant Self Compassion - measured using Self Compassion Scale-Short Form (SCS-SF) | 7 week (Group-A and Group B)
  12-item measure that assesses the ability to demonstrate care and kindness toward oneself, and acceptance of one's own imperfections. Self-compassion is often a focus of mindfulness-based interventions because of the interrelatedness with state mindfulness. Responses will be given using a 5-point Likert scale that ranged from 1 ("Almost never") to 5 ("Almost always"), yielding a total score between 12 and 60, with higher scores indicating greater self-compassion.
Autistic Participant Self Compassion - measured using Self Compassion Scale-Short Form (SCS-SF) | 15 Week (Group-A and Group B)
  12-item measure that assesses the ability to demonstrate care and kindness toward oneself, and acceptance of one's own imperfections. Self-compassion is often a focus of mindfulness-based interventions because of the interrelatedness with state mindfulness. Responses will be given using a 5-point Likert scale that ranged from 1 ("Almost never") to 5 ("Almost always"), yielding a total score between 12 and 60, with higher scores indicating greater self-compassion.
Autistic Participant Self Compassion - measured using Self Compassion Scale-Short Form (SCS-SF) | 22 Week (Group B)
  12-item measure that assesses the ability to demonstrate care and kindness toward oneself, and acceptance of one's own imperfections. Self-compassion is often a focus of mindfulness-based interventions because of the interrelatedness with state mindfulness. Responses will be given using a 5-point Likert scale that ranged from 1 ("Almost never") to 5 ("Almost always"), yielding a total score between 12 and 60, with higher scores indicating greater self-compassion.
Autistic Participant Self Compassion - measured using Self Compassion Scale-Short Form (SCS-SF) | 30 Week (Group B)
  12-item measure that assesses the ability to demonstrate care and kindness toward oneself, and acceptance of one's own imperfections. Self-compassion is often a focus of mindfulness-based interventions because of the interrelatedness with state mindfulness. Responses will be given using a 5-point Likert scale that ranged from 1 ("Almost never") to 5 ("Almost always"), yielding a total score between 12 and 60, with higher scores indicating greater self-compassion.
Autistic Community connectedness (ACC) - measured using Autistic Community Connectedness Measure (ACC) | Baseline/enrolment (Group-A and Group B)
  ACC will be used to measure how connected to the autistic community each participant felt. It comprises of ten statements and is rated on a 6-point Likert scale ranging from 1('strongly disagree') to 6, ('strongly agree'). Total scores range from 10 to 60, with higher scores reflecting greater autistic community connectedness.
Autistic Community connectedness (ACC) - measured using Autistic Community Connectedness Measure (ACC) | 7 week (Group-A and Group B)
  ACC will be used to measure how connected to the autistic community each participant felt. It comprises of ten statements and is rated on a 6-point Likert scale ranging from 1('strongly disagree') to 6, ('strongly agree'). Total scores range from 10 to 60, with higher scores reflecting greater autistic community connectedness.
Autistic Community connectedness (ACC) - measured using Autistic Community Connectedness Measure (ACC) | 15 Week (Group-A and Group B)
  ACC will be used to measure how connected to the autistic community each participant felt. It comprises of ten statements and is rated on a 6-point Likert scale ranging from 1('strongly disagree') to 6, ('strongly agree'). Total scores range from 10 to 60, with higher scores reflecting greater autistic community connectedness.
Autistic Community connectedness (ACC) - measured using Autistic Community Connectedness Measure (ACC) | 22 Week (Group B)
  ACC will be used to measure how connected to the autistic community each participant felt. It comprises of ten statements and is rated on a 6-point Likert scale ranging from 1('strongly disagree') to 6, ('strongly agree'). Total scores range from 10 to 60, with higher scores reflecting greater autistic community connectedness.
Autistic Community connectedness (ACC) - measured using Autistic Community Connectedness Measure (ACC) | 30 Week (Group B)
  ACC will be used to measure how connected to the autistic community each participant felt. It comprises of ten statements and is rated on a 6-point Likert scale ranging from 1('strongly disagree') to 6, ('strongly agree'). Total scores range from 10 to 60, with higher scores reflecting greater autistic community connectedness.
Autistic Participant Satisfaction-measured using Intervention Satisfaction Scale (ISS) | 7 Week (Group-A)
  At the end of virtual mindfulness session. Participants will be asked open-ended questions asking about what they liked best and least about the group, what the biggest challenges they had to attending group meetings, what would make participation easier, and how they would change the group for future participants via an online survey will be distributed at the end of the course with the post-evaluation measures. Participants will be asked to rate some items, how generally true each item was for them using a 5-point scale ranging from 1 ("Never or very rarely true") to 5 ("Very often or always true"), with higher total scores suggesting greater mindfulness (total score range from 0 to 100)
Autistic Participant Satisfaction-measured using Intervention Satisfaction Scale (ISS) | 22 Week (Group B)
  At the end of virtual mindfulness session. Participants will be asked open-ended questions asking about what they liked best and least about the group, what the biggest challenges they had to attending group meetings, what would make participation easier, and how they would change the group for future participants via an online survey will be distributed at the end of the course with the post-evaluation measures.
  Participants will be asked to rate some items, how generally true each item was for them using a 5-point scale ranging from 1 ("Never or very rarely true") to 5 ("Very often or always true"), with higher total scores suggesting greater mindfulness (total score range from 0 to 100).
Autistic Participant reactivity, observing, acting aware, describing, and non-judgment- measured using Five-Facet Mindfulness Questionnaire- Short Form (FFMQ-SF) | Baseline/ enrolment (Group-A and Group B)
  FFMQ-SF will be used to assess five components of mindfulness: observing one's experiences, describing one's experiences, acting with awareness, accepting inner experiences in a nonjudgmental way, and accepting inner experiences without reacting. Participants will be asked to rate how generally true each item was for them using a 5-point scale ranging from 1 ("Never or very rarely true") to 5 ("Very often or always true"), with higher total scores suggesting greater mindfulness (total score range from 24 to 120).
Autistic Participant reactivity, observing, acting aware, describing, and non-judgment- measured using Five-Facet Mindfulness Questionnaire- Short Form (FFMQ-SF) | 7 Week (Group-A and Group B)
  FFMQ-SF will be used to assess five components of mindfulness: observing one's experiences, describing one's experiences, acting with awareness, accepting inner experiences in a nonjudgmental way, and accepting inner experiences without reacting. Participants will be asked to rate how generally true each item was for them using a 5-point scale ranging from 1 ("Never or very rarely true") to 5 ("Very often or always true"), with higher total scores suggesting greater mindfulness (total score range from 24 to 120).
Autistic Participant reactivity, observing, acting aware, describing, and non-judgment- measured using Five-Facet Mindfulness Questionnaire- Short Form (FFMQ-SF) | 15 Week (Group-A and Group B)
  FFMQ-SF will be used to assess five components of mindfulness: observing one's experiences, describing one's experiences, acting with awareness, accepting inner experiences in a nonjudgmental way, and accepting inner experiences without reacting. Participants will be asked to rate how generally true each item was for them using a 5-point scale ranging from 1 ("Never or very rarely true") to 5 ("Very often or always true"), with higher total scores suggesting greater mindfulness (total score range from 24 to 120).
Autistic Participant reactivity, observing, acting aware, describing, and non-judgment- measured using Five-Facet Mindfulness Questionnaire- Short Form (FFMQ-SF) | 22 Week (Group B)
  FFMQ-SF will be used to assess five components of mindfulness: observing one's experiences, describing one's experiences, acting with awareness, accepting inner experiences in a nonjudgmental way, and accepting inner experiences without reacting. Participants will be asked to rate how generally true each item was for them using a 5-point scale ranging from 1 ("Never or very rarely true") to 5 ("Very often or always true"), with higher total scores suggesting greater mindfulness (total score range from 24 to 120).
Autistic Participant reactivity, observing, acting aware, describing, and non-judgment- measured using Five-Facet Mindfulness Questionnaire- Short Form (FFMQ-SF) | 30 Week (Group B)
  FFMQ-SF will be used to assess five components of mindfulness: observing one's experiences, describing one's experiences, acting with awareness, accepting inner experiences in a nonjudgmental way, and accepting inner experiences without reacting. Participants will be asked to rate how generally true each item was for them using a 5-point scale ranging from 1 ("Never or very rarely true") to 5 ("Very often or always true"), with higher total scores suggesting greater mindfulness (total score range from 24 to 120).
Autistic Participant Interoception measured using, Interoception Sensory Questionnaire (ISQ-8) | Baseline (Group-A and Group B)
  ISQ-8 will be used to measure interoception, the ISQ-8 is the first psychometrically validated self-report measure of interoception for autistic adolescents and adults,and is adapted from the ISQ-20. Items are rated on a 5-point likert scale. A higher score indicates more difficulty registering or interpreting interoceptive sensations.
Autistic Participant Interoception measured using, Interoception Sensory Questionnaire (ISQ-8) | 7 Week (Group-A and Group B)
  ISQ-8 will be used to measure interoception, the ISQ-8 is the first psychometrically validated self-report measure of interoception for autistic adolescents and adults,and is adapted from the ISQ-20. Items are rated on a 5-point likert scale. A higher score indicates more difficulty registering or interpreting interoceptive sensations.
Autistic Participant Interoception measured using, Interoception Sensory Questionnaire (ISQ-8) | 15 Week (Group-A and Group B)
  ISQ-8 will be used to measure interoception, the ISQ-8 is the first psychometrically validated self-report measure of interoception for autistic adolescents and adults,and is adapted from the ISQ-20. Items are rated on a 5-point likert scale. A higher score indicates more difficulty registering or interpreting interoceptive sensations.
Autistic Participant Interoception measured using, Interoception Sensory Questionnaire (ISQ-8) | 22 Week (Group B)
  ISQ-8 will be used to measure interoception, the ISQ-8 is the first psychometrically validated self-report measure of interoception for autistic adolescents and adults,and is adapted from the ISQ-20. Items are rated on a 5-point likert scale. A higher score indicates more difficulty registering or interpreting interoceptive sensations.
Autistic Participant Interoception measured using, Interoception Sensory Questionnaire (ISQ-8) | 30 Week (Group B)
  ISQ-8 will be used to measure interoception, the ISQ-8 is the first psychometrically validated self-report measure of interoception for autistic adolescents and adults,and is adapted from the ISQ-20. Items are rated on a 5-point likert scale. A higher score indicates more difficulty registering or interpreting interoceptive sensations.
Autistic participant mental well-being measured using, the Short Warwick-Edinburgh Mental Wellbeing Scale, SWEMWS | Baseline (Group-A and Group B)
  The Short Warwick-Edinburgh Mental Wellbeing Scale, SWEMWS is a 7-item measure of psychological wellbeing. Example items include 'I've been feeling relaxed' and 'I've been interested in new things'. Participants rated items on a 5-point Likert scale ['none of the time' (1) to 'all of the time' (5)]. Scores could range from 14 to 70, and higher scores indicated more positive mental wellbeing.
Autistic participant mental well-being measured using, the Short Warwick-Edinburgh Mental Wellbeing Scale, SWEMWS | 7 Week (Group-A and Group B)
  The Short Warwick-Edinburgh Mental Wellbeing Scale, SWEMWS is a 7-item measure of psychological wellbeing. Example items include 'I've been feeling relaxed' and 'I've been interested in new things'. Participants rated items on a 5-point Likert scale ['none of the time' (1) to 'all of the time' (5)]. Scores could range from 14 to 70, and higher scores indicated more positive mental wellbeing.
Autistic participant mental well-being measured using, the Short Warwick-Edinburgh Mental Wellbeing Scale, SWEMWS | 15 Week (Group-A and Group B)
  The Short Warwick-Edinburgh Mental Wellbeing Scale, SWEMWS is a 7-item measure of psychological wellbeing. Example items include 'I've been feeling relaxed' and 'I've been interested in new things'. Participants rated items on a 5-point Likert scale ['none of the time' (1) to 'all of the time' (5)]. Scores could range from 14 to 70, and higher scores indicated more positive mental wellbeing.
Autistic participant mental well-being measured using, the Short Warwick-Edinburgh Mental Wellbeing Scale, SWEMWS | 22 Week (Group B)
  The Short Warwick-Edinburgh Mental Wellbeing Scale, SWEMWS is a 7-item measure of psychological wellbeing. Example items include 'I've been feeling relaxed' and 'I've been interested in new things'. Participants rated items on a 5-point Likert scale ['none of the time' (1) to 'all of the time' (5)]. Scores could range from 14 to 70, and higher scores indicated more positive mental wellbeing.
Autistic participant mental well-being measured using, the Short Warwick-Edinburgh Mental Wellbeing Scale, SWEMWS | 30 Week (Group B)
  The Short Warwick-Edinburgh Mental Wellbeing Scale, SWEMWS is a 7-item measure of psychological wellbeing. Example items include 'I've been feeling relaxed' and 'I've been interested in new things'. Participants rated items on a 5-point Likert scale ['none of the time' (1) to 'all of the time' (5)]. Scores could range from 14 to 70, and higher scores indicated more positive mental wellbeing.
Follow-up Satisfaction Form | End of the Study
  At the end of the study participants will be asked 8 likert scale close ended questions and 10 open ended questions about what they liked best about the research study what were the biggest challenges they had, what would make participation easier, and what they would change for future participants via online survey at the end of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Yona Lunsky, PhD, Principal Investigator — CAMH
Locations (1):
- CAMH, Toronto, Ontario, Canada